CLINICAL TRIAL: NCT05794542
Title: Cue X as a Treatment for People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Professor Rory O'Connor, Charterhouse Professor of Rehabilitation Medicine, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 321744
Record Dates: First submitted 2022-11-28; First posted 2023-04-03 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Use of Cue X intervention
  Interventions: Device: Cue X

INTERVENTIONS:
Device: Cue X — Cue X is used with augmented (mixed) reality glasses. These glasses are similar to virtual reality glasses except you can see the real world around you with digital images overlain. The Cue X software is used on two existing devices, the Microsoft HoloLens and the Magic Leap.

SUMMARY:
Parkinson's disease is a progressive neurological condition which affects more than 145,000 people in the United Kingdom (UK) today. The main symptoms are tremor (uncontrolled shaking), slowness of movement and difficulty starting movements (termed 'freezing'). Daily exercise is recommended to help with these symptoms.

Rehabilitation can help to maintain a person's balance, ability to walk and help to prevent falls. This can allow people living with Parkinson's to maintain their independence for longer. Rehabilitation is usually carried out at face-to-face appointments in outpatient departments in hospitals.

STROLLL (www.strolll.co) is a company that have created a programme of activities called Cue X, to be used on augmented reality glasses. Augmented reality glasses merge computer generated images and sounds with the real world. Cue X has been created specifically to help people with Parkinson's.

We are aiming to recruit 50 participants through referrals from specialist doctors, nurses and physiotherapists in Leeds Teaching Hospitals National Health Service (NHS) Trust. We will ask these health care professionals to give potential participants an information sheet outlining the project. A more detailed participant information sheet will be sent by post or email to those interested.

There will be an initial hospital appointment where written consent will be asked for and an initial assessment completed. Participants will do a personalised, daily rehabilitation programme using Cue X on augmented reality glasses for 6 weeks at home (monitored remotely by a physiotherapist). A final assessment and review will be done in hospital.

The purpose of this project is to see if people with Parkinson's can use the glasses and do exercises in their own homes. Benefits could include fewer trips to the hospital for appointments and a more engaging way of participating in rehabilitation.

If successful, this could lead further research into this technology as a new way of delivering rehabilitation.

DETAILED DESCRIPTION:
Parkinson's disease is a condition that affects the brain. It is the world's fastest growing neurological condition which affects more than 145,000 people in the United Kingdom (UK) today. No one knows exactly why the condition develops and there is currently no cure for Parkinson's.

The symptoms associated with Parkinson's are usually mild at first, but can become worse over time. The main symptoms are tremor (uncontrolled shaking), slowness of movement and difficulty starting movements. People with Parkinson's often have problems with walking and balance because of these. This can make normal daily activities more difficult.

It is generally recommended that adults are physically active every day to reduce the effects of sedentary behaviour. UK Department of Health and Social Care guidelines for the adult population recommend 150 minutes of moderate intensity physical activity (equivalent to 30 minutes per day, 5 days a week) or 75 minutes of vigorous intensity physical activity a week (gov.uk, 2019). This is no different for people living with Parkinson's. Indeed, people living with Parkinson's are encouraged to engage in a daily exercise programme to maintain their mobility, independence, and quality of life. However, it can be difficult to do exercises because of the disabling symptoms affecting movement. In addition, as gait and balance ability deteriorate, and the fear of falls increases, maintaining an exercise programme becomes more difficult, leading to being less able to do everyday activities and declining quality of life.

Rehabilitation can help people living with Parkinson's to maintain their mobility and independence, as well as assisting in preventing falls. People usually attend outpatient appointments with a specialist rehabilitation team for assessment and are commenced on a treatment programme of advice, exercises and activities. People are reviewed regularly at face-to-face appointments, with treatment plans adjusted as needed.

One particular problem that many people report with their mobility is 'freezing' when walking (termed 'freezing of gait' or FoG). This is when a person stops and is unable to take their next step. Previous research has shown that there are ways to help people when they freeze using visual or auditory cues to provide 'prompts' to take the next step. For example, putting taped lines on the floor to step over, a light on a walking stick or listening to the beat of a metronome. Most of the existing technology relies on someone else being present, carrying a walking aid or the lines being in fixed places on the floor.

A company called Strolll have created a digital programme specifically for people living with Parkinson's. It is called Cue X and is used with augmented (mixed) reality glasses. These glasses are similar to virtual reality glasses except you can see the real world around you with digital images overlain. The Cue X software is used on two existing proprietary devices, the Microsoft HoloLens and the Magic Leap.

The Cue X software used provides access to visual and audio cueing, with the potential for haptic (tactile) cues in the future, in a single wearable device. For each modality, there is a library of games which utilise cues. The cue-assisted gait and balance exercises that underpin the games can be selected to form a rehabilitation programme personalised and adapted to each user aiming to maximise and maintain the positive effect on gait and balance over time. The Cue X supports independent rehabilitation, delivered in augmented reality, to enable people with Parkinson's to participate in exercises without a healthcare professional present, where previously without cueing, walking and balance training would not be possible.

Augmented reality rehabilitation using Cue X has the potential to deliver engaging exercise treatments that can be completed by a person independently at home. This could reduce outpatient face-to-face contact time for staff and patients, while improving experiences, accessibility and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

Age >= 18 years Confirmed Parkinson's diagnosis Under the care of a consultant or Parkinson's specialist nurse in Leeds. Able to walk indoors with or without a walking aid

Exclusion Criteria:

Age < 18 years Skin condition on head or face that prevents wearing the headset Cognitive impairment causing inability to consent Unable to walk at any time Severe visual impairment resulting in inability to see the augmented reality information Epilepsy Mental health condition causing hallucinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L (This is the registered name of the outcome measure) | At 6 weeks: on completion of the intervention
  5-level EuroQoL-5 dimension: health related quality of life assessment

SECONDARY OUTCOMES:
The Parkinson's Disease Questionnaire (PDQ-39) | At 6 weeks: on completion of the intervention
  A Parkinson's Disease-specific health status questionnaire comprising 39 items for health-related quality of life assessment
Lindop Parkinson's Assessment Scale | At 6 weeks: on completion of the intervention
  This is a standardised physiotherapy assessment of a person with Parkinson's disease's ability to move

CONTACTS AND LOCATIONS:
Overall Officials: Rory O'Connor, MD, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No